CLINICAL TRIAL: NCT04068285
Title: Neuromuscular Adaptations to Exercise In Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, GULIN FINDIKOGLU, Associate Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 60116787-0
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Gait, Unsteady; Aerobic Exercise
Keywords: Type 2 diabetes mellitus; exercise; aerobic; interval; continuous; gait
MeSH Terms: conditions — Gait Disorders, Neurologic; Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study has 3 arms.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants wil be making exercise. It is not possible to make participants blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity interval exercise (Active Comparator): Participants with type 2 Diabetes mellitus in High intensity interval exercise (HIIE) group will make aerobic exercise using bicycle at high intensity followed by low intensity periods under observation in the hospital.
  exercise
  Interventions: Other: Aerobic Exercise
- Moderate intensity continuous exercise (Active Comparator): Participants with type 2 Diabetes mellitus in Moderate intensity continuous exercise (MIC) group will make aerobic exercise using bicycle at moderate intensity during the session under observation in the hospital.
  exercise
  Interventions: Other: Aerobic Exercise
- No Intervention: Control group (No Intervention): The participants with type 2 Diabetes mellitus in the control group will make stretching exercise at home

INTERVENTIONS:
Other: Aerobic Exercise — Participants will be making aerobic exercise
  Arms: High intensity interval exercise; Moderate intensity continuous exercise

SUMMARY:
The aim of this study is to compare the effects of high intensity interval exercise and moderate intensity continuous exercise on basic gait parameters in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Volunteers with type 2 diabetes mellitus will be evaluated in terms of any contra-indication that will restrain them from making exercise. 90 male or female volunteers who are suitable in terms of inclusion/exclusion criteria will be invited for the study. Volunteers will be randomly distributed to one of the 3 groups. Each group will contain 30 participants. 1. group will make aerobic exercise which is in the form of high intensity interval exercise 2.group will make aerobic exercise which is in the form of moderate intensity continuous exercise 3. Control group. Exercise groups will be cycling under observation in the hospital setting. Control group will make simple stretching exercises at home. Participants will be requested to complete a 3 months of exercise. They will be evaluated before and at the end of the 3 months of exercise with basic gait parameters such as cadence, gait speed, stride length, percentages of swing phase and stance phase evaluated by a wireless digital miniature gait analysis system.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have type 2 Diabetes mellitus less than 10 years and more than 1 year.
2. Participants must have appropriate medical therapy and diet.
3. Participants must not be treated with insulin.
4. Participants must be exercising less than 210 minutes/ week

Exclusion Criteria:

1. Participants with prominent cardiovascular disease
2. Participants with coronary artery disease
3. Participants with moderate to severe valvular disease
4. Participants with atrial fibrillation
5. Participants with untreated hypertension
6. Participants with congenital heart disease
7. Participants with retinopathy
8. Participants with neuropathy
9. Participants with macro albuminuria
10. Participants with cerebrovascular disease
11. Participants with ejection fraction less than 40
12. Participants with body mass index greater than 35.
13. Participants with prominent ischemic changes in EKG at rest or during exercise.
14. Participants with cigarette or alcohol addiction
15. Participants on drugs that interferes with body fat distribution (such as insulin, thiazolidinediones

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
walking speed | 12 weeks
  change in walking speed in m/s

CONTACTS AND LOCATIONS:
Overall Officials: Gulin Findikoglu, Assoc Prof, Principal Investigator — Pamukkale University,Medical Faculty, PMR Department
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No